CLINICAL TRIAL: NCT02583061
Title: Toronto Gestational Glucose Tolerance Cohort
Status: Recruiting | Type: Observational
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 01-0318-E
Record Dates: First submitted 2015-10-20; First posted 2015-10-21 (Estimated); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes, Gestational Diabetes, Pre-diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes, Gestational; Glucose Intolerance | interventions — Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: There is no intervention. An exposure of interest is glucose tolerance status in pregnancy

SUMMARY:
In this prospective observational cohort study, women representing the full spectrum of gestational glucose tolerance status are undergoing longitudinal cardiometabolic characterization at regular intervals in the years after the index pregnancy.

DETAILED DESCRIPTION:
In this prospective observational cohort study, women reflecting the full spectrum of glucose tolerance in pregnancy (from gestational diabetes mellitus (GDM) to lesser degrees of gestational glucose intolerance to those with completely normal glucose tolerance) are being recruited in late 2nd trimester. This cohort of women thus carries a broad range of risk for the future development of type 2 diabetes (T2DM) and cardiovascular disease. At regular intervals in the years after the index pregnancy, this cohort of women is undergoing serial cardiometabolic characterization, including assessment of glucose tolerance, beta-cell function and insulin sensitivity. The longitudinal changes over time in this cohort should provide insight into the early pathophysiology and natural history of T2DM and cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women

Exclusion Criteria:

* Pre-existing diabetes before the index pregnancy

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of pregnant women across the full spectrum of gestational glucose tolerance
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2003-09; Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Glucose tolerance status | 10 years after pregnancy
  Glucose tolerance is assessed on oral glucose tolerance test

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Retnakaran, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada